CLINICAL TRIAL: NCT03396952
Title: Prostaglandin Inhibition and Programmed Cell Death Protein 1 (PD-1)/Cytotoxic T-lymphocyte-Associated Protein 4 (CTLA4) Blockade in Melanoma
Brief Title: Prostaglandin Inhibition and Immune Checkpoint Blockade in Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17854; NCI-2017-02441 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Results first posted 2021-06-10 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-09

CONDITIONS: Stage III Cutaneous Melanoma; Stage IIIA Cutaneous Melanoma; Stage IIIB Cutaneous Melanoma; Stage IIIC Cutaneous Melanoma; Stage IV Cutaneous Melanoma
MeSH Terms: conditions — Melanoma | interventions — Aspirin; Ipilimumab; CTLA-4 Antigen; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, ipilimumab, aspirin) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1, ipilimumab IV over 60 minutes on day 1 for courses 1-4, and aspirin PO BID (orally, twice a day) on days 1-21. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Aspirin; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Aspirin — Given PO
  Other Names: Acetylsalicylic Acid (ASA); Aspergum; Ecotrin; Empirin; Entericin; Extren; Measurin
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab, ipilimumab, and aspirin work in treating patients with melanoma that has spread to other places in the body or cannot be removed by surgery. Monoclonal antibodies, such as pembrolizumab and ipilimumab, may interfere with the ability of tumor cells to grow and spread. Aspirin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving pembrolizumab, ipilimumab, and aspirin may work better in treating patients with melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the overall response rate (ORR) by week 12 in patients with stage III unresectable/stage IV melanoma.

SECONDARY OBJECTIVES:

I. To determine the median progression free survival, overall survival, and toxicity profile of the combination of ipilimumab, pembrolizumab and high dose aspirin in patients with stage III unresectable/IV melanoma.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1, ipilimumab IV over 60 minutes on day 1 for courses 1-4, and aspirin orally (PO) twice daily (BID) on days 1-21. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed melanoma that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Leukocytes >= 3,000/microliter (mcL)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Total bilirubin =< 1.5 X institutional upper limit
* Aspartate aminotransferase (AST) [serum glutamic-oxaloacetic transaminase (SGOT)] =< 2.5 X institutional upper limit of normal
* Alanine aminotransferase (ALT) [serum glutamate pyruvate transaminase (SGPT)] =< 2.5 X institutional upper limit of normal
* Creatinine =< 1.5 X upper limit of normal (ULN)
* Women of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study drug; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Women of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 120 days after the last dose of study medication; Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Men of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy; Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Ability to understand a written informed consent document, and the willingness to sign it

Exclusion Criteria:

* Any mental or physical condition or disease or past medical history that mitigates against following the protocol
* History of active autoimmune diseases such as but not limited to Crohn?s disease, ulcerative colitis, Sjogren's syndrome, requiring active immune suppression; patient may have hay fever or controlled asthma
* Any solid organ transplant or bone marrow transplant
* Any other disseminated malignancy. Exceptions include: localized prostate cancer, basal or squamous cell skin cancer, localized cervical cancer, and localized breast cancer.
* Uncontrolled central nervous system (CNS) metastasis; patients with CNS metastasis can be eligible if definitively treated with radiotherapy or surgery
* Any coexistent medical condition interfering with drug absorption
* History of gastritis or malabsorption syndrome or aspirin intolerance or allergy
* Live vaccination within the last 30 days
* History of multiple sclerosis, type 1 diabetes mellitus (DM) or Guillain-Barre syndrome
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil Daud, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of Califonia, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Pembrolizumab, Ipilimumab, Aspirin): Patients receive pembrolizumab IV over 30 minutes on day 1, ipilimumab IV over 60 minutes on day 1 for courses 1-4, and aspirin orally, twice a day (PO BID) on days 1-21. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Aspirin: Given orally (PO)
  Ipilimumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Ipilimumab, Aspirin)
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Ipilimumab, Aspirin)
Number analyzed (Participants) | 27
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 3
  40-49 years old | 3
  50-59 years old | 3
  60-69 years old | 8
  70-79 years old | 7
  80-89 years old | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Defined as the proportion of subjects for whom the best overall response at week 12 is confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST). Point estimates of ORR and 95% confidence intervals will be provided. Only participants with confirmed response are included in this analysis.
Time Frame: Up to 12 weeks
Population: Only participants with confirmed response are included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Pembrolizumab, Ipilimumab, Aspirin)
Number analyzed (Participants) | 23
proportion of participants | 0.522 [0.330 to 0.708]

2. Secondary Outcome: Number of Participants With Reported Treatment-related Adverse Events
Description: Number of participants with reported treatment-related adverse events defined as having an attribution of definite, possible, and probable according to Common Terminology Criteria for Adverse Events (CTCAE) version 4 will be reported.
Time Frame: Within 30 days after last dose of study drug, up to 3 years
Measure: Number; unit: particpants
Arm/Group | Treatment (Pembrolizumab, Ipilimumab, Aspirin)
Number analyzed (Participants) | 27
particpants | 5

3. Secondary Outcome: Proportion of Participants With Progression-free Survival (PFS) at 6 Months
Description: PFS at 6 months is defined as the proportion of subjects alive and progression-free 6 months (182 days) after study day 1.
Time Frame: Up to 6 months (182 days)
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Pembrolizumab, Ipilimumab, Aspirin)
Number analyzed (Participants) | 27
proportion of participants | 0.566 [0.336 to 0.74]

4. Secondary Outcome: Median Duration of PFS
Description: Duration of PFS is defined as the time from the study day 1 to the earlier of disease progression or death due to any cause. The analysis of PFS will include only objective progression events per RECIST and clinical progression determined by the investigator may not be considered disease progression. The median duration of PFS will be estimated using the Kaplan-Meier methods with the associated 95% confidence interval.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Ipilimumab, Aspirin)
Number analyzed (Participants) | 27
months | 7.6 [4.9 to 11.0]

5. Secondary Outcome: Median Overall Survival (OS)
Description: Duration of OS is defined as the time from study day 1 to death due to any cause. For subjects who are alive at the time of data cutoff or are permanently lost to follow-up, duration of OS will be right censored at the date the subject was last known to be alive. The median duration of OS will be estimated using the Kaplan-Meier methods with the associated 95% confidence interval.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Ipilimumab, Aspirin)
Number analyzed (Participants) | 27
months | 8.9 [5.0 to 11.3]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Treatment (Pembrolizumab, Ipilimumab, Aspirin)
All-Cause Mortality (participants affected / at risk) | 4/27
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Ipilimumab, Aspirin) (N=27)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Ipilimumab, Aspirin) (N=27)
Abdominal pain (Gastrointestinal disorders) | 11 (14)
Diarrhea (Gastrointestinal disorders) | 10 (19)
Abdominal distension (Gastrointestinal disorders) | 9 (13)
Nausea (Gastrointestinal disorders) | 9 (10)
Constipation (Gastrointestinal disorders) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 17 (19)
Fever (General disorders) | 6 (6)
Pain (General disorders) | 4 (6)
Non-cardiac chest pain (General disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 8 (8)
Hypothyroidism (Endocrine disorders) | 6 (8)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Headache (Nervous system disorders) | 10 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Serum amylase increased (Investigations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2)
Lipase increased (Investigations) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Eye disorders - Other (Eye disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT03396952/Prot_SAP_000.pdf